CLINICAL TRIAL: NCT03319693
Title: Molecular Characterization of Primary Mucosal Melanoma
Acronym: MELMUQ
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA16108*
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Mucosal Melanoma
MeSH Terms: interventions — Genetic Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mucosal melanoma: Incident Mucosal melanoma in the Champagne-Ardenne region 2004-2014
  Interventions: Genetic: Somatic Genetic

INTERVENTIONS:
Genetic: Somatic Genetic — NGS analysis

SUMMARY:
Primary mucosal melanomas (MPM) are rarer than cutaneous melanomas, but also more severe. They are usually refractory to conventional approaches, regularly excluded from major therapeutic programs and not sensitive to new targeted therapies orphans. " The identification of therapeutic targets and accessibility to existing, developing or future targeted therapies improves the survival of patients with MPM.

The principal goal is to describe, using a large panel of genes, the prevalence of major mutations in a cohort of MPMs based on the population of a French region.

ELIGIBILITY:
Inclusion criteria:

* Incident Mucosal melanoma in the Champagne-Ardenne region 2004-2014

Exclusion criteria:

* Cutaneous melanoma
* Uveal melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MPM
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
The frequency of main mutations identified using the NGS panel | Day 0
  NGS panel

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France